CLINICAL TRIAL: NCT06790485
Title: In-Vivo Validation of Novel Diagnostic Devices Versus Visual ICDAS-II Criteria in Detection of Early Occlusal Caries
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Abdel Fattah Mahmoud Edrees, Assistant Professor of Conservative Dentistry, Cairo University
Other Study IDs: 24-058
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Dental Caries (Diagnosis)
MeSH Terms: conditions — Dental Caries; Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient with initial occlusal caries

SUMMARY:
The diagnosis of non-cavitated occlusal caries is considered problematic and still a challenge for dental professionals. It affects 60-90% of schoolchildren and adults.Clinically, caries commonly is performed by methods of visual examination and subjective assessments of, translucency, color and dental hardness, as well as by means of radiographic imaging. These methods, however, show low sensitivity for occlusal caries detection.Some of these methods are light based fluorescence devices taking the advantages of the fluorescence properties of the hard tissues of the tooth as there is a difference in fluorescence observed in sound and demineralized dental tissues.Other methods based on electrical impedance has been used. These devices aimed to employ the AC Impedance Spectroscopy Technique (ACIST) In order to record variations in mineral density throughout the tooth, not just the surface, ACIST sends a low amplitude microamp current from the sensor tip contact through the pulp, dentin, and enamel.Hence, a diagnostic accuracy study control trial is to be held to evaluate the Clinical performance of quantitative light fluorescence based device (Vistacam Proof) and impedance spectroscopy based device (CariescanPRO) in comparison with the visual examination and digital radiography in detection of initial pits and fissures caries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 21 to 50 years.

  * Patient at least has one posterior pits and fissure occlusal caries.
  * No gender restriction
  * Co-operative patients who signed the informed consent.
  * Good general health
  * Acceptable oral health

Exclusion Criteria:

* Pregnancy.

  * Disabilities.
  * Systemic disease or severe medical complications.
  * Allergic history concerning methacrylate.
  * Rampant caries.
  * Heavy smoking.
  * Xerostomia.
  * Lack of compliance.
  * Evidence of severe bruxism, clenching, or temporomandibular joint disorders

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited by researcher according to the eligibility criteria from clinic of conservative dentistry department in Faculty of Dentistry in The British University in Egypt, where there is a continuous and high patient flow
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
primary occlusal caries | 1 week
  posterior tooth with occlusal discoloration

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Other, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edrees A, Hassanein O, Shaalan O, Yassen A. Accuracy of high definition near infrared transillumination camera in detection of hidden proximal caries. J Clin Exp Dent. 2023 Jan 1;15(1):e1-e8. doi: 10.4317/jced.59413. eCollection 2023 Jan. PMID 36755680